CLINICAL TRIAL: NCT06368492
Title: The Impact of Psilocybin on Pain in Fibromyalgia Patients: a Multicentre Trial.
Brief Title: The Impact of Psilocybin on Pain in Fibromyalgia Patients
Acronym: PsiloFM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P137; 2021-002909-10 (EudraCT Number); NL78008.068.21 (Other: METC azM/Maastricht University)
Record Dates: First submitted 2023-10-31; First posted 2024-04-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; psychedelics; psilocybin; chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, within-subjects, placebo-controlled design.
Masking Description: Blinding will be handled by one of the study pharmacies and order and allocation of the treatment to each participant will be completely randomized. This setup ensures that neither the participant nor the experimenter running the test day will be aware of the contents of the capsule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient group (Experimental): Each participant will receive 2 different doses of psilocybin (5mg and 10mg) and a matching placebo on three separate occasions.
  Interventions: Drug: Psilocybin; Behavioral: Hypnosis script

INTERVENTIONS:
Drug: Psilocybin — Each participant will receive 2 different doses of psilocybin (5mg and 10mg) and a matching placebo on three separate occasions.
Behavioral: Hypnosis script — All participants will receive a brief hypnotic induction aimed at producing analgesia before the second administration of CPT

SUMMARY:
Rationale: Recent evidence shows that Lysergic Acid Diethylamide (LSD), even when administered in low, non-hallucinogenic doses, can produce analgesic effects and improve pain tolerance in a sample of healthy volunteers. Such results complement what was already observed with other serotonergic psychedelics such as psilocybin: survey studies and case series indicate that its use may lead to improvements in chronic pain conditions such as migraines, cluster headaches and phantom limb pain even at low, non-psychedelic doses. These effects have however not yet been investigated and confirmed in clinical populations under controlled experimental conditions.

Fibromyalgia (FM) is a chronic condition characterised by widespread pain, hyperalgesia, anxiety, disturbed sleep patterns, impaired cognitive functioning and comorbid mood disorders. Most suggested therapies are only associated with small improvements in pain ratings and quality of life. Currently, there is no data concerning the effectiveness of serotonergic psychedelics in improving pain ratings in fibromyalgia patients.

Objective: The present study will explore the effects that the administration of a placebo and 2 low psilocybin doses (5 mg or 10 mg) will have on pain perception in a group of fibromyalgia patients.

Study design: The present study uses a double-blind, randomized, placebo-controlled design. All participants will receive a placebo and 2 doses of psilocybin (5 mg or 10 mg) and will undergo the Cold Pressor Test (CPT) and the Pain Pressure Threshold Task (PPT) o test its analgesic effects.

DETAILED DESCRIPTION:
Rationale: Recent evidence shows that Lysergic Acid Diethylamide (LSD), even when administered in low, non-hallucinogenic doses, can produce analgesic effects and improve pain tolerance in a sample of healthy volunteers. Such results complement what was already observed with other serotonergic psychedelics such as psilocybin: survey studies and case series indicate that its use may lead to improvements in chronic pain conditions such as migraines, cluster headaches and phantom limb pain even at low, non-psychedelic doses. These effects have however not yet been investigated and confirmed in clinical populations under controlled experimental conditions.

Fibromyalgia (FM) is a chronic condition characterised by widespread pain, hyperalgesia, anxiety, disturbed sleep patterns, impaired cognitive functioning and comorbid mood disorders. It has high direct and indirect costs and it is considered challenging to treat. Most suggested therapies, in fact, are only associated with small improvements in pain ratings and quality of life. Currently, there is no data concerning the effectiveness of serotonergic psychedelics in improving pain ratings in fibromyalgia patients.

Objective: The present study will explore the effects that the administration of a placebo and 2 low psilocybin doses (5 mg or 10 mg) will have on pain perception in a group of fibromyalgia patients.

Study design: The present study uses a double-blind, randomized, placebo-controlled design. All participants will receive a placebo and 2 doses of psilocybin (5 mg or 10 mg) and will undergo the Cold Pressor Test (CPT) and the Pain Pressure Threshold Task (PPT) o test its analgesic effects.

Study population: 35 fibromyalgia patients aged 18 to 65 years. Intervention: Placebo, 5 mg or 10 mg of psilocybin in randomized order. Main study parameters/endpoints: Primary outcomes will be subjective and objective measures of pain perception. Secondary measures will assess the effects that placebo and psilocybin will have on mood, cognition and psychedelic experience. Finally, participants will take part to an additional CPT after receiving hypnotic suggestions of analgesia to test whether such intervention may moderate pain ratings of individuals who took small doses of psilocybin.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants will visit the research lab 5 times during 5 weeks. Before the first study day, subjects will come for a screening visit during which they will also be familiarized with tests and study procedures. This includes a medical screening by a licensed physician (medical history review, laboratory screening, electrocardiogram recording). The study visits will consist of taking the study treatment (5 mg or 10 mg of psilocybin or placebo), taking part to the experimental tasks, taking blood samples, completing computer tasks and filling out questionnaires. Finally, participants will take part to a final online visit to administer post-study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Normal weight, body mass index (weight/height2) between 18 and 28 kg/m2
* Fulfilment of the American College of Rheumatology criteria for FM diagnosis (43)
* A minimum Numeric Rating Scale (numeric rating scale) pain score of 5 out of 10
* Proficient knowledge of the Dutch or English language
* Written Informed Consent
* Understanding the procedures and the risks associated with the study
* No regular use of psychotropic medication such as opiates, antidepressants, muscle relaxants, anticonvulsants, sleep aids, benzodiazepines. Non pharmacological regimens will be allowed along 1 rescue therapy such as acetaminophen ≤4,000 mg/day, ibuprofen ≤1,200 mg/day, naproxen ≤660 mg/day, or ketoprofen ≤75 mg/day. Use of paracetamol (PCM) and non-steroidal anti-inflammatory drugs (NSAIDS) will be allowed and monitored.
* Willingness to refrain from taking psychoactive substances during the study.
* Willingness to drink only alcohol-free liquids and no coffee, black or green tea, or energy drinks after midnight of the evening before the study session, as well as during the study days
* Willingness not to drive a traffic vehicle or to operate machines within 24 h after substance administration

Exclusion Criteria:

* Presence of any other painful condition such as inflammatory rheumatic diseases, migraines or headaches and of other chronic or acute medical conditions
* Presence or history of any other psychiatric condition such as primary major depressive disorder, anxiety disorders or substance use disorder as determined by the medical questionnaire, drug questionnaire and medical examination
* Previous experience of serious side effects to psychedelic drugs (anxiety or panic attacks)
* Tobacco smoking (>20 per day)
* Excessive drinking (>20 alcoholic consumptions per week)
* Psychotic disorder in first-degree relatives
* Pregnancy or lactation
* Hypertension (diastolic > 90 mmHg; systolic > 140 mmHg)
* History of cardiac dysfunctions (arrhythmia, ischemic heart disease…)
* For women: no use of a reliable contraceptive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ischemic Pain perception | 1.5, 2.5 and 4 hours after administration
  Pain tolerance (seconds) in the Cold Pressor Task
Pressure-evoked Pain perception | 1.5 and 4 hours after administration
  Pain threshold (kPa) in the Pressure Pain Threshold
Self-reported pain | 1.5, 2.5 and 4 hours after administration
  Painfulness Visual Analogue Scale (0: no pain; 10 worst pain)

SECONDARY OUTCOMES:
Subjective effects: psychedelic phenomenology | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5 and 6 hours after administration
  5 Dimensions of altered states of consciousness (5D-ASC)
Subjective effects: mood | Baseline, 1, 2, 3, and 5 hours after administration
  Profile of mood states (POMS)
Subjective effects: intensity of effects | Baseline, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5 and 6 hours after administration
  Intensity of effects Visual Analogue Scale (VAS) (0: not under the influence; 10: very much under the influence)
Subjective effects: Ego dissolution | 6 hours after administration
  Ego Dissolution Inventory(EDI)
Subjective effects: Dissociation | Baseline and 6 hours after administration
  Clinical Administered Dissociative States Scale (CADSS)
Psychiatric symptoms | Baseline and 6 hours after administration
  Brief Symptom Inventory (BSI)
Cognitive performance | 1.5 and 4 hours after administration
  Digit Symbol Substitution Test (DSST) - time to complete in seconds and number of errors
Vigilance | 1.5 and 4 hours after administration
  Psychomotor Vigilance Task (PVT) - number of attention lapses
Empathy | 1 hour after administration
  Multifaceted Empathy Test (MET) - emotion recognition accuracy (right answers/wrong answers)
Creativity | 2.5 hours after administration
  Alternate Use Test (AUT) - Fluency and Originality, Flexibility, and Elaboration scores
Creativity | 2 hours after administration
  Story Writing
Autobiographical memory | 2.5 hours after administration
  Autobiographical Memory Test (AMT)
Autobiographical memory | Study baseline and 1 week after last experimental session
  Autobiographical Recollection Test (ART)
Treatment expectancy | Study baseline
  Credibility/Expectancy Questionnaire (CEQ)
Treatment expectancy | Study baseline
  Treatment Expectations in Chronic Pain (TEC)
Fibromyalgia-related pain | Baseline and 1 week after each experimental session
  o Fibromyalgia Impact Questionnaire (FIQ)
Personality | Baseline and 1 week after last experimental session
  Big Five Inventory (BFI)
Absorption | Baseline and 1 week after the experimental session
  Modified Tellegen Absorption Scale (MODTAS)
Interpersonal Reactivity | Baseline and 1 week after last experimental session
  Interpersonal Reactivity Index (IRI)
Depression | Baseline
  o Beck Depression Inventory - II (BDI-II)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes G. Ramaekers, PhD, Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Maastricht University, Maastricht, Limburg
  - Leiden University Medical Center, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellanos JP, Woolley C, Bruno KA, Zeidan F, Halberstadt A, Furnish T. Chronic pain and psychedelics: a review and proposed mechanism of action. Reg Anesth Pain Med. 2020 Jul;45(7):486-494. doi: 10.1136/rapm-2020-101273. Epub 2020 May 4. PMID 32371500

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT06368492/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT06368492/ICF_001.pdf